CLINICAL TRIAL: NCT03704610
Title: Efficacy of Remission-induction Regimen With Infliximab for Severe Extrathoracic Sarcoidosis (EFIRTES STUDY)
Brief Title: Efficacy of Remission-induction Regimen With Infliximab for Severe Extrathoracic Sarcoidosis (EFIRTES)
Acronym: EFIRTES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P141205J; 2017-001809-32 (EudraCT Number)
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-10

CONDITIONS: Extrathoracic Sarcoidosis
Keywords: sarcoidosis; extra-thoracic; infliximab
MeSH Terms: conditions — Sarcoidosis | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the two first infusions will be blinded. Treatment will be prepared by local pharmacies. The pharmacist will receive a fax with the treatment to prepare (infliximab or placebo). The placebo will be an injectable solution of 0.9% sodium chloride equivalent to the one used for infliximab reconstitution. Both treatments will be presented in an infusion bag. After reconstitution and dilution, infliximab solution is clear and limpid, similar to 0.9% sodium chloride solution.
  At week 6, after evaluation of ePOST score, unblinding process will be done. All the patients will receive infliximab treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INFLIXIMAB (Experimental): Infliximab 5 mg/kg D1-D15, then infliximab every 4 weeks W6-W10-W14
  Interventions: Drug: Infliximab
- Placebo (Other): placebo injection D1-D15 then infliximab 5 mg/kg W6-W8-W12-W16-W20
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — An initial period with 2 injections with infliximab allowing the determination of the primary criteria Then an extension with infliximab with 3 supplementary perfusions
  Arms: INFLIXIMAB
Drug: Placebo — An initial period with 2 injections with placebo allowing the determination of the primary criteria Then an extension with infliximab with 5 supplementary perfusions
  Arms: Placebo

SUMMARY:
The present study was designed to assess the efficacy of infliximab in a 2-period study :

* An initial period with comparison of infliximab versus placebo and allowing the determination of the primary criteria
* Then an extension period in which the 2 arms will receive infliximab (in the placebo group : 5 perfusions and in the experimental group 3 supplemental perfusions). Finally, the 2 groups will receive 5 injections of infliximab There is little evidence in the literature of when and how infliximab should be administered in sarcoidosis. We hypothesized, from our personal experience in 30 cases (18 of which were reported in a retrospective trial (14), that infliximab would have a very quick activity. So it appeared reasonable to evaluate the primary criterion at 6 weeks after initiation of the treatment.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystemic granulomatous disease of unknown cause . Sarcoidosis is chronic and progressive in 25 % of the patients. Although mediastinal lymph nodes and lung are the most frequently sites affected, extrathoracic localizations may occur. In particular, cardiac or neurological localizations are frequently associated with a chronic disease, with subsequent morbidity and mortality. Such patients require long term therapy to avoid organ dysfunction which may occur with fibrosis.

If cyclophosphamide remains the "historical" treatment to treat resistant sarcoidosis, it can present serious adverse effects such as infections and gonadic toxicity which may be a problem in young people. As infliximab has demonstrated a real efficacy in resistant sarcoidosis, we challenged that it could be a valuable option for resistant extra-thoracic sarcoidosis.

The population studied will be the patients with clinical and radiological presentation concordant with sarcoidosis

This study is a phase 3, randomized, controlled, parallel group trial, designed to assess the efficacy of infliximab in a 2-period study :

In the first part, patients will be randomly assigned in a 1:1 ratio to receive either infliximab or placebo. Both patients and investigators will be blind regarding study treatment. Concomitantly, patients will be treated with usual care (i.e. steroids at the dose of 0.5 mg/kg/d with a program of tapering dose).

In the second open-labelled part, all the patients will receive infliximab treatment, steroids tapering regimen and low-dose methotrexate left to the investigator choice or, in case of contra-indication, azathioprine.

Finally, the 2 groups will receive 5 injections of infliximab

Infliximab will be used at a dose of 5 mg/kg at D1,D15 then every 4 weeks because in our experience, extrathoracic severe localization require such dosage and may be resistant to the low dosage (3 mg/kg). This dosage is also the dose usually recommended for extra-thoracic localizations.

Disease activity and ePOST score will be evaluated at the inclusion, W6 and after 5 injections (2 weeks after W20 for placebo group or W14 for experimental group). Severity assessment score (ePOST score) will be assessed by the physician in charge of the patient. This score reflects the sarcoidosis activity in 17 organs and has been validated in previous studies.

Remission at week 6 will be defined as: Percentage of patients who have a severity assessment score (ePOST score) inferior to 1 in all organs and absence of hypercalcemia at W6, whatever the corticosteroid dosage received.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological presentation confirming sarcoidosis
* Presence of non caseating granuloma in at least one organ
* Presence of at least one extrathoracic localization, including hypercalcemia
* Exclusion of other causes of granuloma
* Presence of serious organ involvement or relapse/apparition of a new localization despite a first-line immunosuppressive drug
* Age superior or equal to 18 years

Exclusion Criteria:

* Pregnancy or breast feeding or women in age of pregnancy without efficient contraception
* Patients with multiple sclerosis
* Patients with prior history of any cancer in the 5 years before inclusion (except for cutaneous basocellular cancers),
* Patients with a history of hypersensitivity to infliximab to other murine proteins, or to any of the excipients
* Patients with untreated tuberculosis or current other severe infections such as sepsis, abscesses, and opportunistic infections• Patients with moderate or severe heart failure (NYHA class III/IV)
* Concurrent vaccination with live vaccines during therapy
* Inability to understand information about the protocol
* Adult subject under legal protection or unable to consent.
* No informed consent
* Absence of affiliation to National French social security system
* Patients with severe renal failure, severe hepatic impairment, hepatocellular insufficiency, chronic respiratory insufficiency, risk of angle closure glaucoma, risk of urinary retention related to urethroprostatic disorders, certain evolving viral diseases (including hepatitis, herpes, varicella, zoster), psychotic states still not controlled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients | week 6
  who have a severity assessment score (ePOST score) inferior to 1 in all organs and absence of hypercalcemia at W6, whatever the corticosteroid dosage received

SECONDARY OUTCOMES:
Percentage of patients | week 16 for experimental arm ; week 22 for control arm
  who will have completed the steroid tapering regimen, will have a severity assessment score (ePOST score) < 1 in all organs, absence of hypercalcemia, had not have a relapse or any reason for treatment failure
Mean variation in severity assessment score measured by extrapulmonary Physician Organ Severity Tool (ePOST) | Week 6
  ePOST score will be assessed by the physician in charge of the patient. This score reflects the sarcoidosis activity in 17 organs and has been validated in previous studies : Skin, Peripheral lymph nodes, Eyes, Liver, Spleen, Central nervous system, Peripheral nervous system, Parotid/salivary glands, Bone marrow, Ear, Nose, Throat, Cardiac, Renal, Bone/joint, Muscle, Gastrointestinal. For each organ, a score will : 0 as Not affected, 1 as Slight, 2 as Mild, 3 as Moderate, 4 as Moderate to severe, 5 as Severe and 6 as Very severe. Total score is the sum of score in each organ.
Pulmonary sarcoidosis involvement | Week 6
  Pulmonary sarcoidosis involvement will be assessed by the physician in charge of the patient rated as: 0 as Not affected, 1 as Slight, 2 as Mild, 3 as Moderate, 4 as Moderate to severe, 5 as Severe and 6 as Very severe.
Pulmonary sarcoidosis involvement 2 weeks after the 5th injection | week 16 for experimental arm ; week 22 for control arm
  Pulmonary sarcoidosis involvement will be assessed by the physician in charge of the patient rated as: 0 as Not affected, 1 as Slight, 2 as Mild, 3 as Moderate, 4 as Moderate to severe, 5 as Severe and 6 as Very severe.
Severity assessment score measured by ePOST 2 weeks after the 5th injection | week 16 for experimental arm ; week 22 for control arm
  ePOST score will be assessed by the physician in charge of the patient. This score reflects the sarcoidosis activity in 17 organs and has been validated in previous studies : Skin, Peripheral lymph nodes, Eyes, Liver, Spleen, Central nervous system, Peripheral nervous system, Parotid/salivary glands, Bone marrow, Ear, Nose, Throat, Cardiac, Renal, Bone/joint, Muscle, Gastrointestinal. For each organ, a score will : 0 as Not affected, 1 as Slight, 2 as Mild, 3 as Moderate, 4 as Moderate to severe, 5 as Severe and 6 as Very severe. Total score is the sum of score in each organ
Mean variation in the severity assessment score measured by ePOST from 1st injection (W0 or W6) to 2 weeks after the 5th injection | week 16 for experimental arm ; week 22 for control arm
  ePOST score will be assessed by the physician in charge of the patient. This score reflects the sarcoidosis activity in 17 organs and has been validated in previous studies : Skin, Peripheral lymph nodes, Eyes, Liver, Spleen, Central nervous system, Peripheral nervous system, Parotid/salivary glands, Bone marrow, Ear, Nose, Throat, Cardiac, Renal, Bone/joint, Muscle, Gastrointestinal. For each organ, a score will : 0 as Not affected, 1 as Slight, 2 as Mild, 3 as Moderate, 4 as Moderate to severe, 5 as Severe and 6 as Very severe. Total score is the sum of score in each organ.
Mean variation of quality of life measured by SF-36 | Week 6
  The SF-36 questionnaire is a quality of life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. Score from 0 to 100.
Mean variation of fatigue, measured by the Fatigue Scale (FAS) | Week 6
  The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue
Mean variation of quality of life measured by SF-36 | week 16 for experimental arm ; week 22 for control arm
  The SF-36 questionnaire is a quality of life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. Score from 0 to 100.
Mean variation of fatigue, measured by the Fatigue Scale (FAS) | week 16 for experimental arm ; week 22 for control arm
  The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue
Rate of relapses | week 16 for experimental arm ; week 22 for control arm
  A relapse will be defined by the apparition of a new localization or a majoration of the severity assessment score from the previous assessment in at least one organ among the 17 studied in the ePOST score, after a previous 1 point or more decrease without hypercalcemia.

CONTACTS AND LOCATIONS:
Overall Officials: Fleur COHEN AUBART, MCU-PH, Study Director — APHP - Hôpital Pitié-Salpêtriere, Paris,France
Locations (10):
- France (10):
  - Hopital Avicenne - service de pnaumologie, Bobigny
  - Hopital Henri Mondor- service de Médecine Interne, Créteil
  - Hopital Claude Huriez- service de Médecine Interne, Lille
  - Hopital de la Croix Rousse- service de Médecine Interne, Lyon
  - Hopital de la Timone- service de Médecine Internne, Marseille
  - CHU Hotel Dieu - service de Médecine Interne, Nantes
  - GH la Pitié Salpêtrière. Service de Médecine interne, Paris
  - Hopital BICHAT - Médecine Interne, Paris
  - Hopital Bichat- service de pneumologie, Paris
  - Nouvel Hopital Civil- service de Médecine Interne, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.